CLINICAL TRIAL: NCT03411187
Title: Study on the Application of Convenient Foot-control Exhaust Method in Endoscopic Thyroidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bo Wang,MD (Other)
Responsible Party: Sponsor-Investigator, Bo Wang,MD, Clinical Professor, Fujian Medical University
Organization: Fujian Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: exhaust
Record Dates: First submitted 2018-01-19; First posted 2018-01-26 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Thyroid Cancer; Papillary Thyroid Carcinoma; Thyroidectomy; Endoscopy
Keywords: Endoscopy; Thyroidectomy; Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Cancer, Papillary

STUDY DESIGN:
Intervention Model Description: This study is a prospective randomized controlled study to select a continuous case of thyroid surgery in the fujian medical university union hospital from January 2017 to June 2017.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- foot-control exhaust group (Active Comparator): The foot-control exhaust group used of the Pressure adjustable foot-control method by the way of adjustable Pressure to intermittent exhaust
  Interventions: Device: used of the Pressure adjustable foot-control method
- direct exhaust group (Placebo Comparator): direct exhaust group exhaust through the Trocar hole.and without use of the Pressure adjustable foot-control method
  Interventions: Device: direct exhaust

INTERVENTIONS:
Device: used of the Pressure adjustable foot-control method — Whether The Pressure adjustable foot-control method is used.
  Arms: foot-control exhaust group
Device: direct exhaust — direct exhaust through the trocar.
  Arms: direct exhaust group

SUMMARY:
Endoscopic thyroidectomy developed rapidly in recent years, and the most popular surgical approach was endoscopic thyroidectomy by bilateral areola approach, but some operative steps was required optimization. One of the most annoying problem was the smog blurring endoscopic lens during surgery. The researcher summarized a set of convenient foot-control exhaust method and carried out this prospective study.

DETAILED DESCRIPTION:
The patients with papillary thyroid microcarcinoma were included according to the inclusive criteria and randomly divided them into two groups (foot-control exhaust group and direct exhaust group). The foot-control exhaust group used the foot-control exhaust method by the way of adjustable Pressure to intermittent exhaust, while direct exhaust group exhaust through the Trocar hole. Comparison of operation time, times of wiping the endoscopic lens, volume of postoperative drainage, and number of identified parathyroid gland between two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with maximum tumor diameter ≤1 cm;
2. patients without lateral neck lymph node metastases;
3. patients without distant metastases;
4. patients who only needed unilateral surgery following the guidelines;
5. patients with strong cosmetic requirement.

Exclusion criteria:

1. Patients with maximum tumor diameter >1 cm;
2. patients who needed complement total thyroidectomy according to the guidelines, including tumor extrathyroidal extension as well as large amount of neck lymph node metastases and distant metastases;
3. patients without cosmetic requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Flap separation time | 1 day after surgery
  Flap separation time was acquired from endoscopic video was the period from endoscopy into the body to building up operation space.
Glandular excision time | 1 day after surgery
  Glandular excision time was defined from incising cervical white line to removing Berry ligament.
Central lymph node dissection time | 1 day after surgery
  Central lymph node dissection time: was from separating central lymph node to the specimen removed.

SECONDARY OUTCOMES:
Times of wiping lens | 1 day after surgery
  Times of wiping lens calculated from endoscopic video after operation was defined the times of wiping lens from endoscopy into the body to central lymph node removed.
Volume of intraoperative blood loss | 1 day after surgery
  Volume of intraoperative blood loss was estimated the volume of intraoperative blood loss.
Volume of Postoperative drainage | 1 day，2 day，3 day after surgery
  Volume of Postoperative drainage was accurately calculated the total volume while the drainage tube removed after operation.
The number of identifying parathyroid glands | 1 day after surgery
  The number of identifying parathyroid glands was evaluated at postoperation while parathyroid glands was identified during surgery.
Blood PTH level | preoperative, first day after operation, one week after surgery, two months after surgery.
  measurement of PTH level in blood
Blood calcium level | before surgery, the first day after surgery, one week after surgery, two months after surgery.
  to measure the blood calcium level in the blood

CONTACTS AND LOCATIONS:
Locations (1):
- Wen-xin ZHAO, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No